CLINICAL TRIAL: NCT05165238
Title: Impact of a Four-Week Coaching Program on Dietary Habits in Adults With Multiple Sclerosis
Brief Title: Impact Program for Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Brooks C. Wingo, PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 300008553
Record Dates: First submitted 2021-12-17; First posted 2021-12-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coaching program (Experimental): Participants will complete a 4-week coaching program in an on-line group setting. The purpose of the program will be to help participants change dietary behaviors via a small changes approach.
  Interventions: Behavioral: Impact of four week coaching program on dietary habits

INTERVENTIONS:
Behavioral: Impact of four week coaching program on dietary habits — A registered dietitian will provide dietary coaching via online groups to participants.

SUMMARY:
The purpose of this study is to explore the effects of a four week diet coaching program on pain, fatigue, mood, and dietary habits among adults with multiple sclerosis.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is the most common chronic disabling central nervous system (CNS) disease in young adults, affecting 1 in 1,000 people in Western countries. Disproportionate and unpredictable impacts of co-morbid health conditions enhances the needs for comprehensive MS management and wellness strategies.

However, comprehensive care is limited, forcing many people to neglect critical aspects of their wellness. This creates a profound need for health and wellness programs that provide education, connection, and activation.

Research shows a consistent need for more access to reliable information regarding symptoms, management, access to healthcare professionals, and rehabilitation. There is also a primary unmet need for more information on exercise, nutrition, insurance, transportation, and employment.

People living with MS often receive more information from advocacy organizations than their MS nurse or neurologist. Decreased access to healthcare professionals since the COVID-19 pandemic has heightened the need for credible information from organizations like Can Do MS. Over the past year, Can Do MS has seen significant growth in virtual program attendance, with participant identifying "learning new information" as a critical objective.

A multipronged approach utilizing auditory, visual, and kinesthetic learning styles is the preferred method for delivering information. There is also a need to appeal to multiple sensory channels through complimentary mediums (e.g. video, audio, written materials, tactile activities).

We will study the effects of the four week coaching program on dietary patterns in MS patients. This will be done through surveys the participants will complete through Qulatrics.

ELIGIBILITY:
Inclusion Criteria:

All participants will be adults ages 18 to 65 diagnosed with any form of MS. Caregivers are also invited to attend the program if they would like to. No restrictions will be made based on sex, gender or other condition.

Exclusion Criteria:

* If the subjects are outside of the age range they will not be able to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Diet quality | end of intervention (4 weeks)
  Diet quality will be measured via 4 day food journal
Diet quality | 3 months post intervention
  Diet quality will be measured via 4 day food journal

CONTACTS AND LOCATIONS:
Overall Officials: Brooks Wingo, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No